CLINICAL TRIAL: NCT02814513
Title: Feasibility of the ANDAGO System in Pediatric Neurorehabilitation: Bridging the Gap From Treadmill-based to Over-ground Walking
Brief Title: Feasibility of the ANDAGO System in Pediatric Neurorehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huub van Hedel (Other)
Responsible Party: Sponsor-Investigator, Huub van Hedel, PD Dr., University Children's Hospital, Zurich
Organization: University Children's Hospital, Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ANDAGO
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Central Motor Disorders; Orthopedic Disorders
Keywords: Children; Adolescents
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ANDAGO (Experimental): ANDAGO
  Interventions: Device: ANDAGO

INTERVENTIONS:
Device: ANDAGO — Feasibility: the researchers will examine technical features as well as patient-related aspects, safety and operability of the device during static (standing) and dynamic (walking) tasks.
  Other Names: ANDAGO-1
Device: ANDAGO — Differences in static and dynamic tasks when standing/walking in the ANDAGO or when being supervised by a therapist/walking with regular walking aids.
  Other Names: ANDAGO-2
Device: ANDAGO — Investigate the handling of the ANDAGO. Patients will have time to practice with the device and the researchers will evaluate improvements in static/dynamic task performance with the ANDAGO.
  Other Names: ANDAGO-3
Device: ANDAGO — Determine which patients (characterized by demographics and neurological, cognitive and functional status) can improve their handling with the ANDAGO (i.e. whether patients can improve relatively quickly (i.e. 30 minutes of practice time) in dynamic tasks).
  Other Names: ANDAGO-4
Device: ANDAGO — To investigate how well healthy age- and gender matched children can perform the dynamic tasks (obstacle and precision course) and compare these results to those obtained in patients.
  Other Names: ANDAGO-5

SUMMARY:
In this feasibility study, the researchers would like to investigate whether it is feasible to apply the ANDAGO V2.0, a new mobile robot for body-weight supported gait training (developed by Hocoma AG) to children and adolescents undergoing neurorehabilitation. The investigators will explore several outcomes and will compare some outcomes between the children and adolescents when they walk in the ANDAGO or with their regular walking aids.

DETAILED DESCRIPTION:
Background and Rationale:

Children with neurological diagnoses including congenital or acquired brain lesions often have impaired lower extremity function limiting the independence in daily life activities. Achieving the ability to stand and walk independently is mentioned by most children and their parents as the highest priority for the neurorehabilitation process. Robotic gait therapy can deliver high-dosage (i.e. number of practice movements) and high-intensive (i.e. number of movements per unit time) training interventions to complement conventional treatments. Nevertheless, there is a gap between treadmill-based gait training and free walking. HocomaAG (Volketswil) developed a new mobile robot for body-weight supported gait training. ANDAGO will bridge this gap while offering a safe and functional environment for patients. Now, the researchers would like to investigate whether it is feasible to apply this prototype to children and adolescents undergoing neurorehabilitation.

Objective(s):

As the device has not been applied in a pediatric rehabilitation setting yet, the researchers want to investigate:

* Feasibility: the investigators will examine technical features as well as patient-related aspects, safety and operability of the device during static (standing) and dynamic (walking) tasks.
* Differences in static and dynamic tasks when standing/walking in the ANDAGO or when being supervised by a therapist.
* Investigate the handling of the ANDAGO. Patients will have time to practice with the device and Background and Rationale:

Children with neurological diagnoses including congenital or acquired brain lesions often have impaired lower extremity function limiting the independence in daily life activities. Achieving the ability to stand and walk independently is mentioned by most children and their parents as the highest priority for the neurorehabilitation process. Robotic gait therapy can deliver high-dosage (i.e. number of practice movements) and high-intensive (i.e. number of movements per unit time) training interventions to complement conventional treatments. Nevertheless, there is a gap between treadmill-based gait training and free walking. HocomaAG (Volketswil) developed a new mobile robot for body-weight supported gait training. ANDAGO will bridge this gap while offering a safe and functional environment for patients. Now, the researchers would like to investigate whether it is feasible to apply this prototype to children and adolescents undergoing neurorehabilitation.

Objective(s):

As the device has not been applied in a pediatric rehabilitation setting yet, the researchers want to investigate:

* Feasibility: the investigators will examine technical features as well as patient-related aspects, safety and operability of the device during static (standing) and dynamic (walking) tasks.
* Differences in static and dynamic tasks when standing/walking in the ANDAGO or when being supervised by a therapist.
* Investigate the handling of the ANDAGO. Patients will have time to practice with the device and the researchers will evaluate improvements in static/dynamic task performance with the ANDAGO.
* Determine which patients (characterized by demographics and neurological, cognitive and functional status) can improve their handling with the ANDAGO.
* To investigate how well healthy age- and gender matched children can perform the dynamic tasks (obstacle and precision course).

Outcome(s):

Feasibility: outcomes focus on the applicability of the ANDAGO according to therapists' and patients' feedback. The questionnaire includes questions on satisfaction with operability, comfort, safety and the handling of the device, the harnesses and the control panel.

Furthermore the researchers will investigate the precision of the symmetric unloading system with the help of a digital weight scale that the patient steps onto.

The researchers further investigate static balance with a Kistler force plate (Center of Pressure parameters) and time and accuracy of walking with and without the ANDAGO when performing an obstacle and precision course. The investigators will record outcomes like time required to perform the tasks, gait quality with the Edinburgh Visual Gait Score and smoothness of walking with Shimmer sensors, and walking precision with a GoPro camera.

Finally, the researchers assess various characteristics and functional and cognitive outcomes of the patients to correlate these measures with performance and handling of the ANDAGO.

The investigators do not apply any invasive measures and assure that the testing procedures will be limited to keep the burden for the participants acceptable.

Study design:

Open label feasibility study investigating the applicability, safety and handling of the ANDAGO system. Two appointments will be planned for each child within a 48 hour window in order to avoid possible functional improvements due to other therapies. One additional appointment might be planned for clinical, functional or neurological tests that are normally part of our clinical routines. Healthy participants will be appointed only once.

Inclusion/Exclusion criteria:

Children and adolescents from our Rehabilitation Centre, aged between 5 and 18 years, will be included in this project. The investigators expect to recruit 30 participants with central motor disorders or orthopaedic disorders including lower extremity impairments.

Further inclusion criteria are: 1) patients larger than 135 cm, 2) capability to understand and follow simple verbal commands, 3) ability to initiate steps.

The exclusion criteria are: 1) bone fragility of the lower extremities, 2) inability to maintain upright position and lack of head control, 3) uncontrolled hip, knee or ankle instability, 4) elevated risk of seizure, 5) lower extremity contractions (knee > 20°, hip > 20°), 6) presence of skin lesions in areas of contact with the harness support or on feet, 7) implantation of baclofen pump, heart pacemaker or cerebral shunt, 8) cognitive deficit limiting communication of pain or discomfort, 9) limited compliance or aggressive behaviour, 10) any surgical correction or botulinum toxic injection in the lower extremities in the last two months.

Healthy children and adolescents should have no cardiovascular, neurological or musculoskeletal diagnoses.

Measurements and procedures:

Clinical assessments will be performed by therapists to assess the child's functional status regarding muscle strength, selective joint control, spasticity, gait ability and cognitive function.

All exercises will be performed with and without the ANDAGO in a randomized order by each participant.

At the beginning of the first appointment, a standing exercise on a Kistler's force plate will be done. Afterwards the dynamic part of the exercise will be conducted. Participants have to walk along a given path and perform a precision course, followed by an obstacle course. During the second appointment, the participant practices with the ANDAGO and then performs the same obstacle and precision course. Improvements will be objectified by reduced time needed, lower number of prevented falls, higher precision, better gait quality, improved smoothness of walking etc. During the measurements, the children walk with self-selected speed (maximum velocity is 2.1 km/h) and individually adjusted body weight unloading.

Study Product / Intervention:

The ANDAGO V2.0 is a new device. It consists of a stable walking frame and allows a patient to walk with reduced body-weight and without falling over-ground.

Control Intervention (if applicable):

This is a feasibility study, not an RCT; for some tests, the researchers investigate differences in the children's gait capacity when walking with the ANDAGO or without or differences between healthy children and children undergoing neuro-orthopaedic rehabilitation.

Number of Participants with Rationale:

According to the literature, feasibility studies interested in discovering usability for early prototypes are considered valid when including 3-20 participants (Macefield 2008). Due to our heterogeneous patient groups and the potential of some drop-outs, the investigators aim to recruit 30 patients (and an equal number of healthy age- and gender matched controls). These numbers should also be sufficient to detect tendencies of differences within patients (performing static and dynamic tasks with versus without ANDAGO, or improving their handling) or between patients and healthy controls (i.e. differences in the performance of the dynamic tasks between these groups).

Study Duration:

June 2016 - February 2017.

Study Centre(s):

Monocentric study: Rehabilitation Center Affoltern am Albis

Statistical Considerations:

This is not an RCT; therefore there is no primary hypothesis and an accompanying sample size calculation. Depending on the distribution of the data, parametric or non-parametric analyses (e.g. paired-t-test or Wilcoxon signed-rank test for within group differences and t-test or Mann-Whitney U tests for between group comparisons) will be performed. The investigators will correct for multiple comparisons (e.g. Bonferroni correction). Pearson's or Spearman correlations coefficients will be calculated between demographic characteristics and clinical measures versus measures indicating improved handling.

GCP Statement:

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements. will evaluate improvements in static/dynamic task performance with the ANDAGO.

* Determine which patients (characterized by demographics and neurological, cognitive and functional status) can improve their handling with the ANDAGO.
* To investigate how well healthy age- and gender matched children can perform the dynamic tasks (obstacle and precision course).

Outcome(s):

Feasibility: outcomes focus on the applicability of the ANDAGO according to therapists' and patients' feedback. The questionnaire includes questions on satisfaction with operability, comfort, safety and the handling of the device, the harnesses and the control panel.

Furthermore the researchers will investigate the precision of the symmetric unloading system with the help of a digital weight scale that the patient steps onto.

The researchers further investigate static balance with a Kistler force plate (Center of Pressure parameters) and time and accuracy of walking with and without the ANDAGO when performing an obstacle and precision course. The investigators will record outcomes like time required to perform the tasks, gait quality with the Edinburgh Visual Gait Score and smoothness of walking with Shimmer sensors, and walking precision with a GoPro camera.

Finally, the researchers assess various characteristics and functional and cognitive outcomes of the patients to correlate these measures with performance and handling of the ANDAGO.

The investigators do not apply any invasive measures and assure that the testing procedures will be limited to keep the burden for the participants acceptable.

Study design:

Open label feasibility study investigating the applicability, safety and handling of the ANDAGO system. Two appointments will be planned for each child within a 48 hour window in order to avoid possible functional improvements due to other therapies. One additional appointment might be planned for clinical, functional or neurological tests that are normally part of our clinical routines. Healthy participants will be appointed only once.

Inclusion/Exclusion criteria:

Children and adolescents from our Rehabilitation Centre, aged between 5 and 18 years, will be included in this project. The investigators expect to recruit 30 participants with central motor disorders or orthopaedic disorders including lower extremity impairments.

Further inclusion criteria are: 1) patients larger than 135 cm, 2) capability to understand and follow simple verbal commands, 3) ability to initiate steps.

The exclusion criteria are: 1) bone fragility of the lower extremities, 2) inability to maintain upright position and lack of head control, 3) uncontrolled hip, knee or ankle instability, 4) elevated risk of seizure, 5) lower extremity contractions (knee > 20°, hip > 20°), 6) presence of skin lesions in areas of contact with the harness support or on feet, 7) implantation of baclofen pump, heart pacemaker or cerebral shunt, 8) cognitive deficit limiting communication of pain or discomfort, 9) limited compliance or aggressive behaviour, 10) any surgical correction or botulinum toxic injection in the lower extremities in the last two months.

Healthy children and adolescents should have no cardiovascular, neurological or musculoskeletal diagnoses.

Measurements and procedures:

Clinical assessments will be performed by therapists to assess the child's functional status regarding muscle strength, selective joint control, spasticity, gait ability and cognitive function.

All exercises will be performed with and without the ANDAGO in a randomized order by each participant.

At the beginning of the first appointment, a standing exercise on a Kistler's force plate will be done. Afterwards the dynamic part of the exercise will be conducted. Participants have to walk along a given path and perform a precision course, followed by an obstacle course. During the second appointment, the participant practices with the ANDAGO and then performs the same obstacle and precision course. Improvements will be objectified by reduced time needed, lower number of prevented falls, higher precision, better gait quality, improved smoothness of walking etc. During the measurements, the children walk with self-selected speed (maximum velocity is 2.1 km/h) and individually adjusted body weight unloading.

Study Product / Intervention:

The ANDAGO V2.0 is a new device. It consists of a stable walking frame and allows a patient to walk with reduced body-weight and without falling over-ground.

Control Intervention (if applicable):

This is a feasibility study, not an RCT; for some tests, the researchers investigate differences in the children's gait capacity when walking with the ANDAGO or without or differences between healthy children and children undergoing neuro-orthopaedic rehabilitation.

Number of Participants with Rationale:

According to the literature, feasibility studies interested in discovering usability for early prototypes are considered valid when including 3-20 participants (Macefield 2008). Due to our heterogeneous patient groups and the potential of some drop-outs, we aim to recruit 30 patients (and an equal number of healthy age- and gender matched controls). These numbers should also be sufficient to detect tendencies of differences within patients (performing static and dynamic tasks with versus without ANDAGO, or improving their handling) or between patients and healthy controls (i.e. differences in the performance of the dynamic tasks between these groups).

Study Duration:

June 2016 - February 2017.

Study Centre(s):

Monocentric study: Rehabilitation Center Affoltern am Albis

Statistical Considerations:

This is not an RCT; therefore there is no primary hypothesis and an accompanying sample size calculation. Depending on the distribution of the data, parametric or non-parametric analyses (e.g. paired-t-test or Wilcoxon signed-rank test for within group differences and t-test or Mann-Whitney U tests for between group comparisons) will be performed. The investigators will correct for multiple comparisons (e.g. Bonferroni correction). Pearson's or Spearman correlations coefficients will be calculated between demographic characteristics and clinical measures versus measures indicating improved handling.

GCP Statement:

This study will be conducted in compliance with the protocol, the current version of the Declaration of Helsinki, the ICH-GCP or ISO EN 14155 (as far as applicable) as well as all national legal and regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

* >1.35 meter
* Neurological diagnosis
* Orthopaedic diagnosis

Exclusion Criteria:

* Surgery or Botox injection of leg muscles during the last 3 months
* Bone fragility (e.g. non-consolidated fractures or osteotomies including craniotomies, osteopenia, osteoporosis or symptoms or indices in the patient history that infer a higher risk of bone density reduction)
* Unstable arthroplasty
* Uncontrolled knee or ankle instability that would still pose a danger despite the BWS (especially lateral instability)
* Lack of head control
* Joint contractures
* Skin lesions (including pressure sores) in areas of contact with harness support or lower extremity loading (feet)
* Sensory impairment in the lower limbs and trunk, especially with reduced pain sensation
* Risk of autonomic dysreflexia (level at or above T6; history of autonomic dysreflexia increases the risk of having a reoccurring episode)
* Recent history or elevated risk of seizures
* Cardiac conditions, e.g. cardiac insufficiency and thoracotomy, uncontrolled orthostatic hypotension or other circulatory problems, vascular disorders of the lower limbs
* Cognitive deficits limiting communication
* Uncooperative or (self-)aggressive behaviour (e.g. transitory psychotic syndrome)
* Mechanical ventilation
* Long-term infusions (e.g. baclofen pump, Sacral Anterior Root Stimulation (SARS), intrathecal pumps…)
* Any medical condition preventing active rehabilitation (e.g. respiratory disease, pregnancy, orthopaedic conditions, psychiatric conditions, infections or inflammatory disorders, osteomyelitis…)

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09-27 (Actual); Study Completion 2016-09-27 (Actual)

PRIMARY OUTCOMES:
ANDAGO-1: Score on the settings questionnaire | up to 24 weeks
  The Settings questionnaire is a self-developed tool, which covers the following areas:
  * Height of suspension
  * amount of unloading left/right
  * handrails
  * size of the harness and cuffs
  * fall Limit
  * Training mode
  * Maximum velocity
  * turning offset
ANDAGO-2: Position in the ANDAGO device | up to 24 weeks
  Can the patient be positioned well in the ANDAGO? If not, what are the causes? This information is collected for general positioning in the device, fitting of harness and leg "cuffs", both with and without unloading. Furthermore it is asked whether positioning is comfortable for the patient (with or without unloading) and whether there were problems in adjusting parameters like patient lift up and down, bodyweight support, unloading uni- or bilateral. Are there problems in getting the child out of the ANDAGO and did situations occur when patient or therapists needed to press the emergency button?
The Edinburgh Visual Gait Score | up to 24 weeks
  The quality of gait pattern of patients will be assessed within ANDAGO and compared to the walking pattern. Video recordings will be made from the patient and scored according to the Edinburgh Visual Gait Score, which proved one of the most valid and reliable assessments to quantify the quality of the walking pattern. The Edinburgh Visual Gait Score is the sum of the 17 items.
ANDAGO-3: Accuracy of bodyweight support | up to 24 weeks
  The ANDAGO might also be used as a safety system enabling patients to train their standing balance. The researchers will instruct patients to shift their weight as far as possible from the right to the left leg and from anterior to posterior, 5 times in the ANDAGO and 5 times under supervision of a therapist. The investigators will document changes in center of pressure parameters (medio-lateral and anterior-posterior direction), subjective feeling of safety (ordinal smiley scale 1-5), number of "falls" and whether the task could actually be performed or not. Furthermore they report whether the ANDAGO might have limited the exercise and whether the therapist had to intervene during the exercise.
ANDAGO-4: Dynamic obstacle task | up to 24 weeks
  Patients will walk in the ANDAGO or with their regular walking aids and perform an obstacle course. Please note, the steps, obstacles etc. are so narrow that the participant in the ANDAGO can step on them, over them, etc., but the ANDAGO can remain on the flat floor. Participants have to step on a higher surface, a ramp, an uneven surface and over an obstacle. The researchers will assess the time to perform the task, the number of "falls" (patients are secured), subjective feeling of safely (smileys ordinal scale 1-5) and whether the task could be accomplished. Furthermore, they assess whether collisions occurred, whether the ANDAGO limited tasks or whether the therapists needed to intervene.
ANDAGO-5: Dynamic precision task | up to 24 weeks
  Participants will walk 10 meters straightforward, walk a right and left turn and turn around their axis, with and without the ANDAGO. Measures are the time needed to perform these tasks, the number of "falls", the number of steps, precision and smoothness (only with ANDAGO), subjective feeling of safety and whether the task could be accomplished or not. Furthermore, the researchers assess whether collisions occurred, whether the ANDAGO limited tasks or whether the therapists needed to intervene.

CONTACTS AND LOCATIONS:
Overall Officials: Hubertus JA van Hedel, PT, PhD, Principal Investigator — Rehabilitation Center for Children and Adolescents, University Children's Hospital Zurich
Locations (1):
- Rehabilitation Center for Children and Adolescents of the University Children's Hospital Zurich, Affoltern am Albis, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided